CLINICAL TRIAL: NCT02544529
Title: Echothiophate Iodide for the Prevention of Progression of Myopia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding available
Sponsor: Danbury Eye Physicians & Surgeons, PC (Other)
Responsible Party: Principal Investigator, Angela Smit, Director of Clinical Research Operations, Danbury Eye Physicians & Surgeons, PC
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: DEPS 001
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2015-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Echothiophate Iodide; Ophthalmic Solutions; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Echothiophate Iodide (Experimental): Echothiophate Iodide 0.03% one drop to each eye three times per week for 18 weeks
  Interventions: Drug: Echothiophate Iodide 0.03% Ophthalmic Solution
- Carboxymethylcellulose Sodium (0.5%) (Placebo Comparator): Carboxymethylcellulose Sodium (0.5%) one drop to each eye three times per week for 18 weeks
  Interventions: Drug: Carboxymethylcellulose Sodium (0.5%)

INTERVENTIONS:
Drug: Echothiophate Iodide 0.03% Ophthalmic Solution — one drop to each eye three times per week for 18 weeks
  Other Names: Phospholine Iodiede 0.03% ophththalmic solution
  Arms: Echothiophate Iodide
Drug: Carboxymethylcellulose Sodium (0.5%) — one drop to each eye three times per week for 18 weeks
  Other Names: Refresh
  Arms: Carboxymethylcellulose Sodium (0.5%)

SUMMARY:
The purpose of this study is to test the hypothesis that myopia progression can be slowed or prevented by low dose Echothiophate Iodide.

DETAILED DESCRIPTION:
This pilot study is designed to establish proof of concept of a method to either slow or stop the progression of myopia in children between the ages of 8 and 15 years by using Echothiophate Iodide eye drops to alter the relationship between focusing (accommodation), eye alignment, and peripheral blurring. Echothiophate Iodide 0.03% eye drops have been used for years for the treatment of accommodative esotropia in children. A prospective double blind randomized study of 33 children with active development of myopia will be divided into a treatment group of 22 and a control group of 11. They will be treated for 18 weeks with four planned visits at 6 week intervals. The progression of myopia will be measured by a determination of the length of the eye (axial length measured by the IOL Master) and cycloplegic refractions. Influencing factors such as corneal changes, lens changes and macular choroidal thickness will be monitored for any significance. If successful, a larger and longer study to slow the rate of myopia with echothiophate iodide will be done in order to decrease the world's incidence of myopia currently at 25-33% in western countries and 85% in Asian countries. This would also reduce the financial burden of glasses and contact lenses as well as decrease the incidence of pathological eye disease due to high myopia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children between 8-15 years of age
* Documentation of progression of myopia within the 12 months prior to enrollment
* Written informed consent/Assent for the study

Exclusion Criteria:

* Any history of retinopathy of prematurity, glaucoma, cataracts, corneal disease, uveitis, manifest strabismus, nystagmus or ocular trauma
* Any history of unstable asthma, diabetes, or juvenile idiopathic arthritis Asthma must be stable for three months prior to enrollment if utilizing oral or inhaled steroids
* Systemic muscarinic agents, steroids, or anticholinesterase agents.
* Benzalkonium chloride preservative allergy.
* Astigmatism >0.75D
* Anisometropia >1.50D
* Pregnancy or a positive pregnancy test at the screening visit.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-06-01 (Estimated); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Cycloplegic Refraction | 12 weeks
  Cycloplegic refraction change after 12 weeks of treatment with drug

SECONDARY OUTCOMES:
Axial Length | 12 weeks
  Change in axial length after 12 weeks of treatment
Choroidal Thickness | 12 weeks
  Change in choroidal thickness after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Mathias, MD, MPH, Principal Investigator — Danbury Eye Physicians & Surgeons, PC
Locations (1):
- Danbury Eye Physicians & Surgeons, PC, Danbury, Connecticut, United States